CLINICAL TRIAL: NCT01507181
Title: Investigating Rapid Anti-Suicidal Ideation Effects of Intravenous (IV) Ketamine in Hospitalized Patients
Brief Title: Ketamine For Suicidal Ideation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James Murrough (Other)
Responsible Party: Sponsor-Investigator, James Murrough, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 10-1589
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Suicidal Ideation
Keywords: suicidal ideation; major depression; treatment resistant; ketamine; glutamate
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major | interventions — Ketamine; N-Methylaspartate; Excitatory Amino Acid Antagonists; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): single dose IV ketamine, .5mg/kg
  Interventions: Drug: Ketamine
- Midazolam (Placebo Comparator): single dose IV midazolam, .45mg/kg
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — single dose IV ketamine, .5mg/kg infused over 40 minutes
  Other Names: N-methyl-D-aspartate (NMDA) glutamate receptor antagonist
  Arms: Ketamine
Drug: Midazolam — single dose IV midazolam, .45mg/kg infused over 40 minutes
  Arms: Midazolam

SUMMARY:
This study will examine the effects of Intravenous (IV) ketamine both in an outpatient population and with subjects on the inpatient unit with suicidal ideation (SI).

DETAILED DESCRIPTION:
Depression is a debilitating disorder that affects 12-20% of population and is among the top five leading causes of burden of disease worldwide (Kruijshaar ME 2005). Suicide associated with depression and other psychiatric disorders is a pervasive public health problem and results in almost one million deaths per year. Unfortunately, current treatments for severe depression have limited efficacy for suicidality, specifically due to the slow time course of change in suicidal thoughts. Recently ketamine, a glutamate-modulating agent, was shown to have antidepressant and anti-suicidal effect in outpatient depressed patients. The proposed study will test the ability of a single sub-anesthetic intravenous (IV) dose of the glutamate NMDA receptor antagonist, ketamine, to provide rapid decrease in suicidal ideation (SI) in patients hospitalized with SI. In this randomized parallel-arm placebo controlled trial, ketamine is compared to midazolam, which is expected to mimic some of the acute subjective effects of ketamine but not have any sustained antidepressant effects.

Specific Aim 1: To determine feasibility and tolerability of a single low-dose IV infusion of ketamine in patients with prominent SI and elevated risk for suicide.

Hypothesis 1: Ketamine administration will be feasible and well tolerated in patients admitted to a psychiatric hospital with SI.

Specific Aim 2: To test the efficacy of a single IV dose of ketamine, compared to an anesthetic control condition (midazolam), to rapidly reduce SI in a controlled hospital setting.

Hypothesis 2: Ketamine will be associated with significant and rapid reductions in SI and depressive symptoms within 24 hours.

This study will test the rapid anti-suicidal effect of a single IV dose of the N-methyl-D-aspartate (NMDA) glutamate receptor antagonist ketamine in suicidality compared with the clinical response to a single IV dose of the short-acting benzodiazepine midazolam. Midazolam is able to induce transient neuropsychiatric effects mimicking ketamine and therefore is expected to protect the integrity of the blind. Participants will continue to receive standard treatment for their psychiatric condition throughout the trial. This unique "proof-of-concept" study in suicidal patients will be conducted over three-year period.

ELIGIBILITY:
Inclusion Criteria:

* English speaking Male or female patients, 18-80 years
* Patients have voluntarily admitted themselves to an inpatient psychiatric unit at MSH or, regarding the outpatient population, have clinically significant suicidal ideation without intent to harm themselves
* Women of childbearing potential must have a negative pregnancy test
* Clinically significant suicidal ideation and score of ≥4 on MADRS item 10 for suicidality
* Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document

Exclusion Criteria:

* Lifetime history of schizophrenia or other primary psychotic disorder
* Current presence of psychotic symptoms
* Lifetime history of a clearly established psychotic episode
* Established diagnosis of Schizoid, Schizotypal or Paranoid personality disorder
* Urine toxicology screen positive for drugs of abuse on admission
* Substance abuse or dependence within the preceding 1 month
* Anticipated discharge within 7 days of study enrollment (for patients in the inpatient arm)
* Women who plan to become pregnant, are pregnant or are breast-feeding
* Concurrent course of electroconvulsive therapy (ECT)
* Any unstable medical illness including hepatic, renal, gastro-enterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG
* The presence of any known or suspected contraindications to midazolam or ketamine including, but not limited to, known allergic reactions to these agents or acute intermittent porphyria
* Uncontrolled hypertension, defined as BP systolic >160 or BP diastolic >100 on medications
* Arrhythmia requiring medication
* Severe coronary artery disease, defined as Canadian Cardiovascular Status III or IV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Murrough JW, Soleimani L, DeWilde KE, Collins KA, Lapidus KA, Iacoviello BM, Lener M, Kautz M, Kim J, Stern JB, Price RB, Perez AM, Brallier JW, Rodriguez GJ, Goodman WK, Iosifescu DV, Charney DS. Ketamine for rapid reduction of suicidal ideation: a randomized controlled trial. Psychol Med. 2015 Dec;45(16):3571-80. doi: 10.1017/S0033291715001506. Epub 2015 Aug 12. PMID 26266877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the inpatient psychiatric service or through an academic outpatient psychiatric clinic. All study treatments were performed at Mount Sinai Hospital between April 2012 and June 2014.
Period: Overall Study
Arm/Group | Ketamine | Midazolam
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Midazolam | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (15.2) | 39.1 (10.6) | 42.4 (13.3)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 4 | 8
History of suicide attempt [Number; unit: participants]
  yes | 6 | 9 | 15
  no | 6 | 3 | 9
BSI score, baseline [Mean (Standard Deviation); unit: units on a scale] — Beck Scale for Suicidal Ideation - Beck Scale is a 21-item self or clinician administered instrumentation used to measure the current intensity of patients' specific attitudes, behaviors and plans to commit suicide. Score range 0-42, with higher score indicating higher intensity.
  units on a scale | 17.5 (7.2) | 17.9 (11.9) | 17.7 (9.7)
MADRS score, baseline [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale - The MADRS is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  units on a scale | 35.2 (6.1) | 34.3 (4.1) | 34.8 (5.1)
Primary Diagnosis [Number; unit: participants]
  MDD | 6 | 7 | 13
  Bipolar disorder | 4 | 3 | 7
  PTSD | 1 | 2 | 3
  BPD | 1 | 0 | 1
Co-occurring disorders [Number; unit: participants]
  MDD | 2 | 2 | 4
  PTSD | 2 | 1 | 3
  BPD | 1 | 0 | 1
  Panic disorder | 3 | 1 | 4
  SAD | 2 | 4 | 6
  OCD | 3 | 3 | 6
  GAD | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Beck Scale for Suicidal Ideation (BSSI)
Description: Change in BSI score at 24 hours following treatment as compared to baseline. Beck Scale is a 21-item self or clinician administered instrumentation used to measure the current intensity of patients' specific attitudes, behaviors and plans to commit suicide. Score range 0-42, with higher score indicating higher intensity.
Time Frame: baseline and 24 hours post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Midazolam: single dose IV midazolam, .045mg/kg
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
units on a scale | 10.8 (8.5) | 14.0 (10.2)
Statistical Analysis 1: Comparison: Ketamine vs Midazolam; Test type: Superiority or Other; p = 0.32, t-test, 2 sided

2. Primary Outcome: Change in Beck Scale for Suicidal Ideation (BSSI)
Description: Change in BSI score at 48 hours following treatment as compared to baseline. Beck Scale is a 21-item self or clinician administered instrumentation used to measure the current intensity of patients' specific attitudes, behaviors and plans to commit suicide. Score range 0-42, with higher score indicating higher intensity.
Time Frame: baseline and 48 hours post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
units on a scale | 8.8 (8.3) | 15.3 (10.9)
Statistical Analysis 1: Comparison: Ketamine vs Midazolam; Test type: Superiority or Other; p = 0.047, t-test, 2 sided

3. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
Time Frame: up to 7 days post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
units on a scale
  24 hours | 19.0 (15.5) | 26.2 (10.8)
  48 hours | 19.3 (13.5) | 28 (12.3)
  72 hours | 20.9 (14.5) | 24.1 (12.2)
  7 days | 21.7 (13.1) | 22.2 (13.1)
Statistical Analysis 1: Comparison: Ketamine vs Midazolam; Test type: Superiority or Other; p = 0.17, ANCOVA — Statistics are calculated by comparing 24-h scores using separate ANCOVAs and controlling for baseline severity

4. Secondary Outcome: Suicidality Item of the MADRS (MADRS-SI)
Description: The MADRS-SI ranges from 0 to 6; a score of 2 corresponds to fleeting, passive SI; a score of 4 indicates that SI is frequent with at least moderate intensity but without specific plans or intention; a score of 6 corresponds to active intention and planning for suicide.
Time Frame: 24 hours post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
units on a scale | 1.8 (1.9) | 3.3 (1.6)

5. Secondary Outcome: The Young Mania Rating Scale (YMRS)
Description: An 11-item questionnaire, used to assess manic symptoms based on the patient's subjective report of his or her clinical condition. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. The scores from each question are added together to form a total score ranging from 0 to 60, with higher scores indicating a greater severity of symptoms.
Time Frame: baseline, 40 minutes post infusion, 240 minutes post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
units on a scale
  baseline | 0.0 (0.0) | 0.1 (0.3)
  40 minutes post infusion | 0.0 (0.0) | 0.3 (0.6)
  240 minutes post infusion | 0.2 (0.6) | 0.2 (0.6)

6. Secondary Outcome: The Brief Psychiatric Rating Scale (BPRS)
Description: The BPRS measures psychomimetic effects with higher scores indicating more severe symptoms (scale range 7 - 49).
Time Frame: baseline, 40 minutes post infusion, and 240 minutes post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
units on a scale
  baseline | 7.7 (1.12) | 7.7 (1.3)
  40 minutes post infusion | 9.9 (3.3) | 7.9 (1.8)
  240 minutes post infusion | 8.1 (1.6) | 7.0 (0.1)

7. Secondary Outcome: The Clinician-Administered Dissociative States Scale (CADSS)
Description: The CADSS measures dissociation with higher scores indicating more severe symptoms (scale range 0 - 92).
Time Frame: baseline, 40 minutes post infusion and 240 minutes post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
units on a scale
  baseline | 1.1 (2.6) | 4.0 (7.0)
  40 minutes post infusion | 17.1 (19.9) | 3.3 (3.1)
  240 minutes post infusion | 1.2 (1.9) | 1.3 (2.6)

8. Secondary Outcome: Patient Rated Inventory of Side Effects (PRISE)
Description: The PRISE assesses the presence of treatment side effects in nine organ/function systems (gastrointestinal, nervous system, heart, eyes/ears, skin, genital/urinary, sleep, sexual functioning, and other). Data reported in in Adverse Events section.
Time Frame: duration of study
Measure: Number; unit: events
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 12
events | 29 | 23

ADVERSE EVENTS:
Arm/Group | Ketamine | Midazolam
Serious Adverse Events (participants affected / at risk) | 5/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=12) | Midazolam (N=12)
Hospitalizations (Psychiatric disorders) | 4 | 0 — Depression
Death (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Cardiopulmonary disorder unrelated to study participation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=12) | Midazolam (N=12)
Headache (Nervous system disorders) | 7 (7) | 3 (3)
Dizziness on standing (Nervous system disorders) | 2 (2) | 3 (3)
Nausea/Vomiting (General disorders) | 1 (1) | 3 (3)
Diarrhea (General disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Poor concentration (General disorders) | 2 (2) | 1 (1)
Poor coordination (Nervous system disorders) | 2 (2) | 0 (0)
General malaise (General disorders) | 2 (2) | 0 (0)
Restlessness (General disorders) | 2 (2) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Frequent urination (Renal and urinary disorders) | 1 (1) | 1 (1)
Difficulty sleeping (General disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size is small, increasing the likelihood of a false negative finding due to limited power. Unknown if the lack of significant separation between the treatment and control conditions at 24 h represents a true null finding or a false negative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes